CLINICAL TRIAL: NCT00184184
Title: Registration of Tobacco, Coffee and Substance Use Among Acutely Admitted Psychiatric Patients
Status: Completed | Type: Observational
Sponsor: Norwegian University of Science and Technology (Other)
Collaborators: St. Olavs Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: GB- TKR 2004
Record Dates: First submitted 2005-09-12; First posted 2005-09-16 (Estimated); Last update posted 2017-03-14 (Actual); Status verified 2017-03

CONDITIONS: Substance Abuse; Tobacco Use Disorder
Keywords: Emergency Services, Psychiatric; Tobacco use cessation; Coffee use cessation; substance use detection; Substance Abuse Detection
MeSH Terms: conditions — Substance-Related Disorders; Tobacco Use Disorder; Tobacco Use Cessation

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
This is a study of the registration of tobacco, coffee and substance abuse among acutely admitted psychiatric patients.

DETAILED DESCRIPTION:
We will include all patients acutely admitted to Østmarka Psychiatric Hospital to register this population's use of coffee, tobacco and substances. We will determine whether this differs from other populations, between diagnoses, age, etc.

We will also compare results of substance in immunologic rapid urine tests taken by the nurse at the hospital with substance in urine tested in laboratory with LC/MS (liquid chromatography/mass spectrometry).

ELIGIBILITY:
Inclusion Criteria:

* All patients acutely admitted to Østmarka Psychiatric Hospital

Exclusion Criteria:

* Dementia
* Serious brain damage

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 262 (Actual)
Dates: Start 2004-10 (Actual); Primary Completion 2005-06 (Actual); Study Completion 2005-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Gunnar Morken, MD, PhD, Principal Investigator — Norwegian ministry of Education and Research
Locations (1):
- Østmarka Psychiatric Department, St. Olavs Hospital, University Hospital of Trondheim, Trondheim, Norway

REFERENCES:
- [Result] Bagoien G, Morken G, Zahlsen K, Aamo T, Spigset O. Evaluation of a urine on-site drugs of abuse screening test in patients admitted to a psychiatric emergency unit. J Clin Psychopharmacol. 2009 Jun;29(3):248-54. doi: 10.1097/JCP.0b013e3181a45e78. PMID 19440078